CLINICAL TRIAL: NCT07166406
Title: Phase III Randomized Trial of IO-Based Systemic Treatment +/- Liver SBRT in Hepatocellular Cancer With Macrovascular Invasion (HELIO-RT)
Brief Title: Testing Immunotherapy With or Without Stereotactic Body Radiation Therapy in Patients With Advanced Liver Cancer, HELIO-RT Trial
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRG-GI012; NCI-2025-05951 (Other: NCI Trial Identifier)
Record Dates: First submitted 2025-09-03; First posted 2025-09-10 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Advanced Hepatocellular Carcinoma; Stage III Hepatocellular Carcinoma AJCC v8; Stage IV Hepatocellular Carcinoma AJCC v8
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — atezolizumab; Immunoglobulin G; Bevacizumab; Specimen Handling; Magnetic Resonance Spectroscopy; X-Rays; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole; tremelimumab; Disulfides; durvalumab; Nivolumab; Ipilimumab; Radiosurgery

STUDY DESIGN:
Intervention Model Description: No Data Available
Masking Description: No Data Available
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Arm 1 treatment A (atezolizumab, bevacizumab) (Active Comparator): Patients receive atezolizumab and bevacizumab IV every 3 weeks in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection, chest CT and CT and/or MRI throughout the study and may also undergo PET/CT prior to registration.
  Interventions: Biological: Atezolizumab; Biological: Bevacizumab; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Other: Questionnaire Administration
- Arm 1 treatment B (tremelimumab, durvalumab) (Active Comparator): Patients receive tremelimumab IV once and durvalumab IV every 4 weeks in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection, chest CT and CT and/or MRI throughout the study and may also undergo PET/CT prior to registration.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Biological: Tremelimumab; Biological: Durvalumab
- Arm 1 treatment C (nivolumab, ipilimumab) (Active Comparator): Patients receive nivolumab and ipilimumab IV every 3 weeks for up to 4 doses followed by nivolumab IV every 4 weeks in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection, chest CT and CT and/or MRI throughout the study and may also undergo PET/CT prior to registration.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Biological: Nivolumab; Drug: Ipilimumab
- Arm 2 treatment A (atezolizumab, bevacizumab, SBRT) (Experimental): Arm 2 treatment A (atezolizumab, bevacizumab, SBRT) Patients undergo liver SBRT QD, QOD, or twice weekly for 5 fractions over up to 3 weeks. Patients also receive atezolizumab and bevacizumab IV every 3 weeks in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection, chest CT and CT and/or MRI throughout the study and may also undergo PET/CT prior to registration.
  Interventions: Biological: Atezolizumab; Biological: Bevacizumab; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Other: Questionnaire Administration
- Arm 2 treatment B (tremelimumab, durvalumab, SBRT) (Experimental): Patients undergo liver SBRT QD, QOD, or twice weekly for 5 fractions over up to 3 weeks. Patients also receive tremelimumab IV once and durvalumab IV every 4 weeks in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection, chest CT and CT and/or MRI throughout the study and may also undergo PET/CT prior to registration.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Biological: Tremelimumab; Biological: Durvalumab; Radiation: Stereotactic Body Radiation Therapy
- Arm 2 treatment C (nivolumab, ipilimumab, SBRT) (Experimental): Patients undergo liver SBRT QD, QOD, or twice weekly for 5 fractions over up to 3 weeks. Patients receive nivolumab and ipilimumab IV every 3 weeks for up to 4 doses followed by nivolumab IV every 4 weeks in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection, chest CT and CT and/or MRI throughout the study and may also undergo PET/CT prior to registration.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Biological: Nivolumab; Drug: Ipilimumab; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Biological: Atezolizumab — Given IV
  Other Names: 1380723-44-3, Atezolizumab (Tecentriq, ATEZOLIZUMAB), Immunoglobulin G1, Anti-CD274 mAb (MPDL3280A), RG7446, RO5541267
  Arms: Arm 1 treatment A (atezolizumab, bevacizumab); Arm 2 treatment A (atezolizumab, bevacizumab, SBRT)
Biological: Bevacizumab — Given IV
  Other Names: 216974-75-3, Bevacizumab (BEVACIZUMAB, bevacizumab), Avastin, Alymsys, Avzivi, Aybintio, Equidacent, Mvasi, Onbevzi, Oyavas, Vegzelma, Zirabev.
  Arms: Arm 1 treatment A (atezolizumab, bevacizumab); Arm 2 treatment A (atezolizumab, bevacizumab, SBRT)
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection, Biological Sample Collection, Biospecimen Collected, Biospecimen Collection, Specimen Collection
Procedure: Computed Tomography — Undergo CT and PET/CT
  Other Names: CAT, CT, CT scan, CAT scan, Computed Axial Tomography, Computed Tomography (CT), Computerized Tomography, Diagnostic CAT Scan, tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance, MRI, MR, MR Imaging, MRI Scan, Magnetic Resonance Imaging (MRI/procedure/scan), Nuclear Magnetic Resonance Imaging (NMR/NMRI), sMRI, Structural MRI, Medical Imaging
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography (PET), PET scan, PET SCAN, positron emission tomography (procedure/scan)
Other: Questionnaire Administration — Ancillary studies
Biological: Tremelimumab — Given IV
  Other Names: 745013-59-6, Anti-CTLA4 Human mAb (CP-675206/CP675), Imjudo, Immunoglobulin G2, Anti-(Human CTLA-4) mAb (Clone 11.2.1 heavy chain, disulfide)
  Arms: Arm 1 treatment B (tremelimumab, durvalumab); Arm 2 treatment B (tremelimumab, durvalumab, SBRT)
Biological: Durvalumab — Given IV
  Other Names: 1428935-60-7, Durvalumab (DURVALUMAB, Imfinzi), Immunoglobulin G1, Anti-B7-H1 mAb (MEDI4736, heavy/kappa-chain disulfide, dimer
  Arms: Arm 1 treatment B (tremelimumab, durvalumab); Arm 2 treatment B (tremelimumab, durvalumab, SBRT)
Biological: Nivolumab — Given IV
  Arms: Arm 1 treatment C (nivolumab, ipilimumab); Arm 2 treatment C (nivolumab, ipilimumab, SBRT)
Drug: Ipilimumab — Given IV
  Other Names: 477202-00-9, Ipilimumab (IPILIMUMAB, Yervoy), Anti-CTLA-4 mAb (BMS-734016, MDX-010/MDX-CTLA4), Ipilimumab biosimilar CS1002
  Arms: Arm 1 treatment C (nivolumab, ipilimumab); Arm 2 treatment C (nivolumab, ipilimumab, SBRT)
Radiation: Stereotactic Body Radiation Therapy — Undergo liver SBRT
  Other Names: Biological Sample Collection, Biological Sample Collection, Biospecimen Collected, Biospecimen Collection, Specimen Collection
  Arms: Arm 2 treatment B (tremelimumab, durvalumab, SBRT); Arm 2 treatment C (nivolumab, ipilimumab, SBRT)
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography (PET), PET scan/PET SCAN, positron emission tomography (procedure/scan)
  Arms: Arm 2 treatment A (atezolizumab, bevacizumab, SBRT)

SUMMARY:
This phase III trial compares the effect immunotherapy (IO) with stereotactic body radiation therapy (SBRT) to IO alone in treating patients with liver cancer (hepatocellular cancer) that may have spread from where it first started to nearby tissue, lymph nodes, or distant parts of the body (advanced). The usual approach is treatment with IO-based drug combinations, such as atezolizumab and bevacizumab, durvalumab and tremelimumab, or ipilimumab and nivolumab. Durvalumab and tremelimumab are monoclonal antibodies that may interfere with the ability of tumor cells to grow and spread. A monoclonal antibody is a type of protein that can bind to certain targets in the body, such as molecules that cause the body to make an immune response (antigens). IO with monoclonal antibodies, such as atezolizumab, nivolumab and ipilimumab, may help the body's immune system attack the tumor, and may interfere with the ability of tumor cells to grow and spread. Bevacizumab is in a class of medications called antiangiogenic agents. It works by stopping the formation of blood vessels that bring oxygen and nutrients to tumor. This may slow the growth and spread of tumor cells. Radiation therapy uses high energy x-rays, particles, or radioactive seeds to kill cancer cells and shrink tumors. SBRT is a type of external radiation therapy that uses special equipment to position a patient and precisely deliver radiation to tumors in the body (except the brain). The total dose of radiation is divided into smaller doses given over several days. This type of radiation therapy helps spare normal tissue. Giving IO with SBRT may be more effective than IO alone in helping patients with advanced hepatocellular cancer live longer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if liver SBRT in combination with IO-based systemic therapy improves survival compared to IO-based systemic therapy alone, in patients with hepatocellular cancer with macrovascular invasion.

SECONDARY OBJECTIVES:

I. To evaluate and compare progression-free survival between treatment arms. II. To evaluate and compare objective response rate between treatment arms. III. To evaluate and compare vascular recanalization between treatment arms. IV. To evaluate and compare biochemical decline in alpha-fetoprotein (AFP) between treatment arms.

V. To evaluate and compare toxicity within and between treatment arms. VI. To evaluate and compare liver decompensation per Child Pugh score between treatment arms.

VII. To evaluate and compare liver decompensation per modified albumin-bilirubin (ALBI) (mALBI) score between treatment arms.

HEALTH-RELATED QUALITY OF LIFE (HRQOL) OBJECTIVES:

I. To compare Functional Assessment of Cancer Therapy-Hepatobiliary (FACT-Hep) total score at 6 months between the treatment arms. (Primary) II. To evaluate and compare quality-adjusted survival using European Quality of Life Five Dimension (EQ-5D) between treatment arms. (Secondary) III. To evaluate FACT-Hep total scores over time between the treatment arms. (Exploratory)

EXPLORATORY OBJECTIVES:

I. Biospecimen collection for future correlative analyses.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM 1: Patients receive 1 of 3 IO-based systemic treatments per physicians decision.

TREATMENT A: Patients receive atezolizumab and bevacizumab intravenously (IV) every 3 weeks in the absence of disease progression or unacceptable toxicity.

TREATMENT B: Patients receive tremelimumab IV once and durvalumab IV every 4 weeks in the absence of disease progression or unacceptable toxicity.

TREATMENT C: Patients receive nivolumab and ipilimumab IV every 3 weeks for up to 4 doses followed by nivolumab IV every 4 weeks in the absence of disease progression or unacceptable toxicity.

ARM 2: Patients receive 1 of 3 IO-based systemic treatments per physicians decision.

TREATMENT A: Patients undergo liver SBRT once daily (QD), once every other day (QOD), or twice weekly for 5 fractions over up to 3 weeks. Patients also receive atezolizumab and bevacizumab IV every 3 weeks in the absence of disease progression or unacceptable toxicity.

TREATMENT B: Patients undergo liver SBRT QD, QOD, or twice weekly for 5 fractions over up to 3 weeks. Patients also receive tremelimumab IV once and durvalumab IV every 4 weeks in the absence of disease progression or unacceptable toxicity.

TREATMENT C: Patients undergo liver SBRT QD, QOD, or twice weekly for 5 fractions over up to 3 weeks. Patients receive nivolumab and ipilimumab IV every 3 weeks for up to 4 doses followed by nivolumab IV every 4 weeks in the absence of disease progression or unacceptable toxicity.

Additionally, patients undergo blood sample collection, chest computed tomography (CT) and CT and/or magnetic resonance imaging (MRI) throughout the study and may also undergo positron emission tomography (PET)/CT prior to registration.

After completion of study treatment, patients are followed every 3 months for 2 years, every 6 months for 3 years then yearly.

ELIGIBILITY:
* PRIOR TO STEP 1 REGISTRATION:
* Diagnosis of hepatocellular carcinoma (HCC) by at least 1 criterion listed below:

  * Pathologically (histologically or cytologically) proven diagnosis of HCC (strongly recommended)
  * Radiographically proven (American Association for the Study of Liver Diseases [AASLD] criteria) diagnosis of HCC by multiphasic MRI and/or CT scan is allowed.
  * For patients with a prior or concurrent malignancy, pathologic confirmation of hepatocellular cancer is required.
* HCC macrovascular invasion, defined as enhancing vascular thrombosis demonstrating arterial enhancement and venous or delayed venous washout on multiphasic MRI and/or CT is required.
* Presence of extrahepatic metastatic disease on CT chest and CT or MRI pelvis, or PET/CT chest/abdomen/pelvis is permitted.
* 5 or fewer discrete intrahepatic parenchymal foci of HCC.
* Total maximal sum of hepatocellular carcinoma tumors, as a single conglomerate, multiple lesions, or infiltrative HCC < 20 cm in total summed diameter.
* No direct primary tumor extension into the stomach, duodenum, small bowel, or large bowel.
* No known fibrolamellar HCC, sarcomatoid HCC, or biphenotypic HCC.
* Child-Pugh class A or B7 liver function.
* Age ≥ 18.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Not pregnant and not nursing

  * Negative urine or serum pregnancy test (in persons of childbearing potential) within 30 days prior to registration. Childbearing potential is defined as any person who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal.
* Absolute neutrophil count (ANC) ≥ 1,500 cells/mm^3.
* Platelets ≥ 60,000 cells/mm^3.
* Hemoglobin ≥ 8g/dl (Note: The use of transfusion or other intervention to achieve hemoglobin [Hgb] ≥ 8g/dl is acceptable).
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 6 x institutional upper limit of normal (ULN).
* Total bilirubin < 4 x institutional ULN.
* Creatinine clearance (CrCL) ≥ 30 mL/min/1.73 m^2 by the Cockcroft-Gault formula.
* For treatment of HCC:

  * Prior surgical resection, transarterial chemoembolization (TACE), and ablation are permitted.
  * No prior systemic therapy or transarterial radioembolization (TARE) for HCC.
  * No history of liver transplantation.
* For prior treatment for any malignancy:

  * Prior systemic therapy for a different cancer is allowable, except for prior immunotherapy.
  * No prior radiotherapy to the region of the study cancer that would result in significant overlap of radiation therapy fields that would lead to excessive cumulative toxicity at the discretion of the investigator.
* No medical contraindication to the standard of care immunotherapy.
* For patients to be treated with atezolizumab/bevacizumab:

  * No history of a gastrointestinal (GI) bleed or other clinically significant bleeding event within 6 months prior to study registration.
* Systemic immunostimulatory agents (including, but not limited to, interferons and interleukin-2 [IL-2]) are prohibited within 4 weeks or five drug elimination half-lives (whichever is longer) prior to registration and during the study period.
* No history of allergic reaction to the systemic therapy agent(s), compounds of similar chemical or biologic composition to the systemic therapy agent(s) (or any of its excipients).
* PRIOR TO STEP 2 RANDOMIZATION:
* Obtain confirmation of payment coverage (insurance or other) for both possible treatment arms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2025-10-07 (Actual); Primary Completion 2029-03-09 (Estimated); Study Completion 2029-03-10 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | From the date of randomization to the date of death or last follow-up, assessed up to 4 years
  Will be estimated by the Kaplan-Meier method (Kaplan 1958). The distributions of the OS estimates between the two arms will be compared using a log-rank test. The Cox regression model will be used to analyze the effects of factors, in addition to treatment, including, but not limited to stratification factors, which may be associated with OS.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From the date of randomization to the date of first PFS failure or last follow-up for patients without a reported PFS event, assessed up to 4 years
  Will be estimated by the Kaplan-Meier method (Kaplan 1958) and estimates between treatment arms will be compared using the log-rank test (Mantel 1966). The Cox proportional hazard regression model will be used to analyze the effects of factors, in addition to treatment, which may be associated with PFS (Cox 1972).
Objective response rate (ORR) | Up to 4 years
  Will be defined as having a complete or partial response. ORR will be compared between treatment arms using a chi-squared test. Duration of response will also be reported.
Vascular recanalization (VR) | Up to 4 years
  Will be defined as having a complete or partial vascular thrombosis response. The VR proportion for each treatment arm will be determined and compared between treatment arms using a chi-squared test. Time to best VR response before progression and duration of VR response will be reported, but no statistical testing will be done.
Incidence of grade >= 4 adverse events (AEs) (Experimental arm | Up to 90 days from randomization
  Will be compared between the treatment arms using a Z-test.
Safety of stereotactic body radiation therapy with immunotherapy-based systemic therapy | Up to 90 days from randomization
  Will be defined as grade >= 4 AEs definitely related to protocol treatment. Will be compared between the treatment arms using a Z-test.
Selected long-term treatment-related toxicity | Up to 18 months after randomization
  Will focus on grade >=4 hepatobiliary or gastrointestinal AEs and any grade 5 AE. The percentage of patients with the above-specified treatment related AEs will be compared between the treatment arms using a Z-test.
Biochemical decline in alpha-fetoprotein (BD-AFP) | Up to 4 years
  Will be defined as a ≥ 20% decrease in AFP from baseline. The BD-AFP proportion for each treatment arm will be determined and compared between treatment arms using a chi-squared test.
Liver decompensation rate per Child Pugh score (LDR-CP) | Up to 4 years
  The LDR-CP proportion for each treatment arm will be determined and compared between treatment arms using a chi-squared test.
Liver decompensation rate per modified albumin-bilirubin (ALBI) score (LDR-mALBI) | Up to 4 years
  The LDR-mALBI proportion for each treatment arm will be determined and compared between treatment arms using a chi-squared test.

OTHER OUTCOMES:
Functional Assessment of Cancer Therapy-Hepatobiliary (FACT-Hep) total score at 6 Months | At baseline, then at 6 months
  Mean FACT-Hep total score will be compared between treatment arms using a t-test, if normality is met, or Wilcoxon rank-sum test if not. Regression modeling will be used to analyze the effects of factors (e.g. stratification factors and other relevant baseline factors), in addition to treatment, that may be associated with 6-month mean FACT-Hep total score. No statistical testing will be done for subscales.
FACT-Hep total score over time | At baseline and at 3, 6, and 12 months from randomization
  A mixed effects model will be used to assess changes over time. Fixed effects will include baseline scores, treatment arm, stratification factors, as well as the interaction between time and treatment. If the interaction between time and treatment is significant at the 0.05 level, t-tests assessing the between arm difference at each timepoint, within the context of the model, will be conducted
Quality-adjusted survival | At baseline and at 3, 6, and 12 months post treatment completion
  The quality-adjusted survival of each treatment will be evaluated and compared using European Quality of Life Five Dimension (EQ-5D) scale, if the primary endpoint supports the primary hypothesis and/or the EQ-5D significantly differs between treatment arms. The EQ-5D is a 2-part self-assessment questionnaire. To examine trade-offs between the survival time and QOL, they will be combined for each patient into a single measurement: quality-adjusted life years (QALY). If (and only if) the primary endpoint hypothesis is substantiated, a quality-adjusted survival analysis will be conducted. QALY is defined by the weighted sum of different time episodes added up to a total quality-adjusted survival time. QALY will be analyzed using the EQ-5D, using a 2-sided alpha=0.025 to adjust for multiple comparisons.

CONTACTS AND LOCATIONS:
Locations (83):
- United States (83):
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Palo Alto Medical Foundation-Fremont, Fremont, California
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center at Glastonbury, Glastonbury, Connecticut
  - Smilow Cancer Hospital Care Center at Greenwich, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Smilow Cancer Hospital-Hamden Care Center, Hamden, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital Care Center at Long Ridge, Stamford, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Grady Health System, Atlanta, Georgia
  - Emory Proton Therapy Center, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Memorial Hospital East, Shiloh, Illinois
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Waukee Clinic, Waukee, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - The Iowa Clinic PC, West Des Moines, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Allegiance Health, Jackson, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Henry Ford Wyandotte Hospital, Wyandotte, Michigan
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Inova Alexandria Hospital, Alexandria, Virginia
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Inova Fair Oaks Hospital, Fairfax, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Inova Loudoun Hospital, Leesburg, Virginia
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin
  - Essentia Health-Hayward Clinic, Hayward, Wisconsin
  - Essentia Health-Spooner Clinic, Spooner, Wisconsin
  - Essentia Health Saint Mary's Hospital - Superior, Superior, Wisconsin

IPD SHARING:
Plan to Share IPD: No